CLINICAL TRIAL: NCT02797288
Title: Clostridioides Difficile and Immune Responses in Acute CDI and Fecal Microbiota Transplant
Brief Title: Immune Response to C.Difficile Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, William Petri, MD, PhD, Vice Chair, Department of Medicine, University of Virginia
Other Study IDs: 18782; R01AI124214-01 (NIH)
Record Dates: First submitted 2016-05-27; First posted 2016-06-13 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Clostridium Difficile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, and Colon biopsies and brushings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute CDI cohort: Hospitalized patients diagnosed with Acute CDI
- FMT cohort: Patients undergoing FMT for recurrent CDI
- Past CDI Control Cohort: Hospitalized patients with past CDI diagnosis without recurrence

SUMMARY:
The protocol aims to address the basic mechanisms of Clostridium difficile pathogenesis by identifying how a Th 17 response impacts severity of C. difficile infection and how Type II immunity protects the gut from Clostridium difficile toxin-induced damage. This could lead to new and effective approaches to the treatment or prevention of Clostridium difficile colitis that act downstream of fecal microbiota transplants (FMT) or next generation probiotics. Successful fecal microbial transplantation will restore protective immunity to recurrent C.difficile infection.

DETAILED DESCRIPTION:
The study includes one cohort of hospitalized patients with acute CDI who may require diagnostic colonoscopy, a second cohort of outpatients with recurrent CDI scheduled for FMT and a third cohort of inpatients with past history of CDI without recurrence.

Blood samples and discarded stool samples for research will be obtained from adult hospitalized patients. Biopsies and brushing samples for research will be obtained from patients requiring diagnostic colonoscopies for clinical care. Follow-up will include phone contact at 60-90 days to determine relapse or mortality in acute CDI patients.

Blood and colonic biopsies and brushing samples will be obtained from patients undergoing FMT for recurrent CDI and again after 60 days from convalescent patients.

Blood and biopsies taken for research purposes at each colonoscopy will be analyzed for: cytokines and chemokines, gene expression analysis, immunohistochemistry and high dimensional flow-cytometry.

ELIGIBILITY:
Inclusion Criteria:

-Acute CDI cohort

* Acute CDI diagnosis including PCR positive fecal samples
* Optional diagnostic colonoscopy for clinical care

FMT cohort

* At least one relapse or recurrence of C. difficile infection
* Eligible for fecal microbiota transplant (FMT)

Past CDI cohort

* Past CDI diagnosis and current PCR negative fecal samples
* Optional diagnostic colonoscopy for clinical care

Exclusion Criteria:

Acute CDI cohort:

* Unwilling to have research biopsies and brushings at time of diagnostic colonoscopy; Unwilling to provide blood and stool samples (discarded stool from UVA lab) for research
* Unwilling to participate in follow-up phone call at 60-90 days
* Concurrent participation in another clinical trial. This exclusion does not apply to participation in IRB-HSR #200046 and non-interventional research studies. Concurrent participation in non-interventional research studies is allowed.
* Clinical contraindication to colonoscopy or conscious sedation
* Pregnancy
* Inability to give informed consent unless a legally authorized representative (LAR) is available
* Incarceration
* HIV infection

FMT cohort:

* Unwilling to have research biopsies and brushings and stool samples at time of colonoscopy with FMT for clinical care and research sigmoidoscopy at Day 60
* Unwilling to provide blood samples for research
* Concurrent participation in another clinical trial This exclusion does not apply to participation in non-interventional research studies. Concurrent participation in non-interventional research studies is allowed.
* Clinical contraindication to sigmoidoscopy or conscious sedation
* Pregnancy
* Inability to give informed consent
* Incarceration
* HIV infection
* Neutropenia (<1000 PMNs/µl blood)

Past CDI Control cohort:

* Unwilling to have research biopsies and brushings at time of diagnostic colonoscopy; Unwilling to provide blood and stool samples (discarded stool from UVA lab) for research
* Concurrent participation in another clinical trial. This exclusion does not apply to participation in IRB-HSR #200046 and non-interventional research studies. Concurrent participation in non-interventional research studies is allowed.
* Clinical contraindication to colonoscopy or conscious sedation
* Pregnancy
* Inability to give informed consent unless a legally authorized representative (LAR) is available
* Incarceration
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute CDI cohort: Hospitalized patients diagnosed with CDI
  FMT cohort: Adult patients receiving fecal transplant for recurrent CDI identified from the University of Virginia complicated Clostridium difficile clinic
  Past CDI Control cohort: Hospitalized patients with past CDI without recurrence
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Adaptive immune response | 0-60 days post enrollment
  Assessment of adaptive immunity including Th1, Th2 and TH17 immune response

SECONDARY OUTCOMES:
Changes in gut health | 0-60 days post enrollment
  Association of biomarkers in stool and biopsy specimens with CDI outcome
Gene expression of immune cells in colon | 0-60 days post enrollment
  Profiling colonic gene expression and mucosal immune pathways in CDI
Microbiome | 0-60 days post enrollment
  Tissue 16s rDNA
Immunohistochemistry | 0-60 days post enrollment
  Changes in mucosal immunity following FMT
Antibody response to C. difficile infection | 0-60 days post enrollment
  IgG and IgA to C. difficile antigens in plasma and stool
High dimensional flow-cytometry | 0-60 days post enrollment
  Profiling of immune cells in blood and biopsy

CONTACTS AND LOCATIONS:
Overall Officials: William A. Petri, MD,PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreau GB, Tian J, Natale NR, Naz F, Young MK, Nayak U, Tanyuksel M, Rigo I, Madden GR, Abhyankar MM, Hagspiel N, Brovero S, Worthington M, Behm B, Marie C, Petri WA Jr, Ramakrishnan G. Fecal microbiota transplantation promotes type 2 mucosal immune responses with colonic epithelium proliferation in patients with recurrent Clostridioides difficile. JCI Insight. 2025 Nov 18;11(1):e195678. doi: 10.1172/jci.insight.195678. eCollection 2026 Jan 9. PMID 41252206

DOCUMENTS (1):
  • Informed Consent Form (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT02797288/ICF_000.pdf